#### STATISTICAL ANALYSIS PLAN

STUDY TITLE: A Phase 2, Randomized, Double-Blind, Placebo-Controlled

Study to Evaluate the Safety and Efficacy of FG-3019 in

Patients with Idiopathic Pulmonary Fibrosis

PROTOCOL NUMBER: Protocol FGCL-3019-067, Amendment 5.0

**SPONSOR:** FibroGen, Inc.

409 Illinois Street

San Francisco, California 94158 USA

Version Part 2 (Treatment Extension) Final

Release Date: March 14, 2018

#### **CONFIDENTIALITY STATEMENT**

The information contained in this document is confidential and proprietary to FibroGen, Inc. No part of this document or any of the information contained herein may be transmitted, disclosed, shared, reproduced, published or utilized by any persons without prior written authorization by FibroGen, Inc.

## STATISTICAL ANALYSIS PLAN SIGNATURE PAGE

## **Approvals**

I have reviewed and accepted the information in this document to be a true and accurate representation of the Statistical Analysis Plan for analysis of extension data for Study FGCL-3019-067 (Part 2), Extended Treatment Period.

| Initiator: | | |
|------------|-----------------------------------------|-------|
| Signature: | | Date: |
| | Project Statistician,<br>FibroGen, Inc. | |
| Reviewed b | py: | |
| Signature: | | Date: |
| | FibroGen, Inc. | |
| | ribrogen, inc. | |
| Signature: | | Date: |
| | FibroGen, Inc. | |
| Signature: | riorogen, inc. | Date: |
| | FibroGen, Inc. | |

## Signature Significance

The following significance is lent to the signatures on the Approvals page of this document.

| Signatory | Significance |
|---|---|
| Initiator | By signing, the author is attesting that the content of the document is complete and accurate. |
| Reviewer | By signing, the reviewer is attesting that the document's approach and contents are compliant with the study protocol, all appropriate, regulatory requirements, and other significant guidelines. This individual(s) has reviewed the document for accuracy and completeness. |

# Table of Contents

| 1 | INT | RODUCTION | 6 |
|---|---|---|---|
| 2 | Stuc | ly Design (Extended Treatment Period) | 7 |
| | 2.1 | Enrollment to Extended Treatment | 7 |
| | 2.2 | Assessments in Extended Treatment Period | 7 |
| 3 | Stuc | ly Endpoints and Definitions (Extended Treatment Period) | 9 |
| | 3.1 | Study Endpoints | 9 |
| | 3.2 | Definitions of Endpoints in Extended Treatment Period | 9 |
| | 3.2. | 1 Efficacy Endpoints | 9 |
| | 3.2. | 2 Study Drug Exposure and Treatment Compliance | 9 |
| | 3.2. | 3 Adverse Events | 9 |
| | 3.2. | 4 Patient-Exposure-Years | 10 |
| | 3.2. | 5 TEAE and Mortality | 11 |
| 4 | Gen | eral Statistical Considerations | 12 |
| | 4.1 | Analysis Populations | 12 |
| | 4.2 | Handling Dropouts and Missing Data | 12 |
| | 4.3 | Definition of Baseline | 12 |
| | 4.4 | Efficacy Analysis Visit Window | 12 |
| | 4.5 | General Layout | 12 |
| 5 | Stat | istical Analyses | 13 |
| | 5.1 | Subject Disposition | 13 |
| | 5.2 | Protocol Deviations | 13 |
| | 5.3 | Demographic and Baseline Characteristics | 13 |
| | 5.4 | Summary of Prior and Concomitant Medications | 13 |
| | 5.5 | Summary of Study Drug Exposure and Treatment Compliance | 13 |
| | 5.6 | Summary of the Efficacy Data in the Extension Period | 13 |
| | 5.7 | Summary of Safety Data in the Extension Period and Overall Study | 13 |
| | 5.7. | Summary of Treatment Emergent Adverse Events and Mortality | 13 |
| | 5.7. | 2 Summary of Other Safety Data | 13 |
| 6 | Cha | nges from the Protocol | 14 |
| A | ppendi | x. General Specifications for Submission Data | 15 |
| | 1. Stuc | ly Data Tabulation Model (SDTM) | 15 |

| 2 Analysis Data Model | (ADaM) | 18 |
|-----------------------|--------|----|
|-----------------------|--------|----|

#### List of Abbreviations

ADaM Analysis Data Model

AE Adverse event

CM Concomitant medication

CTGF Connective tissue growth factor

ECG Electrocardiogram

EOS End of study

EOT End of treatment

EX Extension

FG-3019 FibroGen-3019 (recombinant human monoclonal antibody)

FVC Forced vital capacity

FVC (L) FVC in litre

FVCpp FVC % predicted

HAHA Human anti-human antibody

HRCT High resolution computed tomography

HRQoL health-related quality of life

ICF Informed consent form

IPF Idiopathic pulmonary fibrosis

PEY Patient exposure years

PK Pharmacokinetic

PRO Patient reported outcome

SAE Serious adverse event

SAP Statistical analysis plan

SGRQ Saint Georges Respiratory Questionnaire

SDTM Study Data Tabulation Model

TEAE Treatment emergent adverse event

## 1 INTRODUCTION

The planned analyses for the Randomized Treatment Period are documented in Part 1 of the Statistical Analysis Plan (SAP) for study FGCL-3019-067: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of FG 3019 in Patients with Idiopathic Pulmonary Fibrosis. This is the part 2 of the SAP, which documents the planned analyses for the Extended Treatment Period. This document is based on the protocol Amendment 5.0 dated 12DEC2016.

In this document, only new definitions and rules will be described; the same definitions and rules described in the Part 1 of the SAP will not be repeated.

## 2 STUDY DESIGN (EXTENDED TREATMENT PERIOD)

#### 2.1 Enrollment to Extended Treatment

### Subjects Enrolled under the Original Protocol and Randomized to FG-3019

All subjects in Arm A whose FVC percent predicted value shows less than 3% absolute decrease from baseline in the Randomized Treatment Period will be offered participation in an Extended Treatment Period. These subjects may continue treatment until FVC percent predicted decreases 3% or more on two consecutive scheduled evaluations compared to the original pre-treatment baseline.

## Subjects Enrolled Under Protocol Amendments and Randomized to FG-3019

All subjects in Arm A whose FVC percent predicted value is greater than the original pretreatment baseline in the Randomized Treatment Period will be offered participation in an Extended Treatment Period and may continue treatment until FVC percent predicted is equal to or less than the pre-treatment baseline on two consecutive scheduled evaluations.

## **Subjects Randomized to Placebo**

All subjects randomized to Placebo (Arm B) will be offered participation in the Extended Treatment Phase for 45 weeks. Placebo subjects in the extension study are treated identically to subjects randomized to FG-3019 in Amendment 1, except for the fact that the baseline for these patients is the time at which they are enrolled into the extension phase (Baseline for Placebo subjects is Week 48 value). Change in FVC percent predicted during the extended treatment phase will be compared to this new baseline. Those subjects whose FVC percent predicted value is either equal to or greater than the new baseline may continue treatment with FG-3019 until FVC percent predicted is equal to or less than the baseline on two consecutive scheduled evaluations.

#### **Subjects in Substudy**

Subjects in substudy are not eligible to enroll into the extended treatment.

#### 2.2 Assessments in Extended Treatment Period

- FVC and FEV1 are assessed at 12-week intervals.
- HRCT scan of the chest is performed at 24-week interval during extension period.
- SGRQ questionnaire is administered at 12-week intervals.
- Electrocardiogram (ECG) is assessed at 24-week intervals.
- Laboratory samples for safety assessments are collected at 6-week intervals.
- Serum and plasma samples for biomarker tests (including CTGF) are collected at 24-week intervals.
- Plasma samples for assessing HAHA are collected prior to dosing on Day 1 of Extension Period and at the End of Study (EOS) safety follow-up.
- Adverse events, concomitant medications, procedures, non-drug therapies, oxygen use are collected from signing ICF through End of Study (EOS).

- Vital signs are measured at every clinical visit. On dosing days, vital signs are measured at pre-, intra-, and post-infusion.
- Physical examination is performed at 6-week intervals.

## 3 STUDY ENDPOINTS AND DEFINITIONS (EXTENDED TREATMENT PERIOD)

### 3.1 Study Endpoints

- Change from baseline in FVC (L) and FVC (% predicted) at each assessed time point
- Change from baseline in fibrosis score by quantitative HRCT at each assessed time point
- Change from baseline in HRQoL at each assessed time point.

## 3.2 Definitions of Endpoints in Extended Treatment Period

### 3.2.1 Efficacy Endpoints

For subjects who were originally randomized to FG-3019, efficacy endpoints are defined as change from the original baseline at study entry. These summaries will enable evaluation of long-term effect.

For subjects who were originally randomized to placebo and rolled over to active in extension, efficacy endpoints are defined as change from baseline as defined as the final assessment during the Randomized Treatment Period. These summaries will enable separate evaluation of effect of active treatment from placebo.

## 3.2.2 Study Drug Exposure and Treatment Compliance

Duration of year 1 exposure = date of last non-zero dose in year 1 – date of first dose +1.

Duration of extended treatment exposure = date last non-zero dose in extension – date of first dose in extension +1.

Duration of entire study treatment exposure = date last non-zero dose in study - date of first dose in study + 1.

Number of infusions is defined as the number of non-zero dose infusions.

Compliance in each treatment year = (# of actual doses administered)/ (# of expected doses) \* 100, where # of expected doses = (last dosing week)/3 + 1. All components in the formula are winthin each treatment year from Day 1 - EX year k to Weeks 45 or EOT in year k.

Overall compliance in entire study = (sum of # of actual doses administered in each treatment year)/ (sum of # of expected doses in each treatment year) \* 100.

#### 3.2.3 Adverse Events

In this SAP Part 2, treatment emergent AE (TEAE) will be defined for (a) the entire study, (b) the Randomized Treatment Period, and (c) the Extended Treatment Period.

TEAE in the Entire Study (TEAE)

TEAEs in the study are defined as <u>new</u> or <u>worsening</u> AEs that occurred in the window of first infusion and within 28 days of the last infusion of study drug, regardless of large gaps of treatment interruption.

TEAE in the Randomized Treatment Period (TEAE-R)

TEAEs during the randomized treatment period are defined as <u>new</u> or <u>worsening</u> AEs that occurred in the window of first dose of infusion of the blinded study drug (FG-3019 or placebo)

(Day 1) and within 28 days of the last infusion of FG-3019/placebo or before the first FG-3019 infusion in the extended treatment period, whichever occurs first.

TEAE in the Extended Treatment Period (TEAE-EX)

TEAEs-EX are defined as <u>new</u> or <u>worsening</u> AEs that occurred in the window of first infusion in Extension and within 28 days of the last infusion in Extension.

Below is an example of the three definitions of TEAE for multiple records of the same AE.

| <b>A</b> E # | Period | Onset | AE | Severity | Serious<br>-ness | Related to study drug? | TEAE | TEAE-R | TEAE-EX |
|---|---|---|---|---|---|---|---|---|---|
| 1 | Year 1 | Screening | Headache | 2 | N | N | N | N | N |
| 2 | Year 1 | Day 2 | Headache | 1 | N | N | N | N | N |
| 3 | Year 1 | Last Year 1<br>dose | Headache | 2 | N | Y | N | N | N |
| 4 | Year 1 | 10 days post<br>last dose | Headache | 3 | Y | N | Y | Y | N |
| 5 | Year 1 | 45 days post<br>last dose | Headache | 4 | Y | N | Y | Y | N |
| 6 | EX | Day 2-EX | Headache | 2 | N | Y | N | N | N |
| 7 | EX-2 | Day 10 EX-<br>2 | Headache | 1 | N | N | N | N | N |
| Consolidated for Entire study summary | | | Headache | 4 | Y | Y | Y | | |
| Consolidated for Year 1 summary | | | Headache | 4 | Y | Y | | Y | |
| Consolidated for Extension summary | | | {none} | NA | NA | NA | | | N |

#### 3.2.4 Patient-Exposure-Years

Patient-Exposure-Years (PEY) is defined as the sum of all subjects' duration of follow-up in years, on FG-3019 or placebo respectively, for the entire study. A subject's duration of follow-up is defined as time from the first dose to the last follow-up recorded in the database. For those

who died, their date of death is the date of last follow-up. For subjects who are randomized to placebo and treated in extension, their last follow-up on placebo is defined as the date prior to Day 1-EX. For other subjects, date recorded on End-of-Study Disposition is the date of last follow-up.

## 3.2.5 TEAE and Mortality

TEAE and mortality will be reported in percentage per total number of subjects exposed.

#### 4 GENERAL STATISTICAL CONSIDERATIONS

Efficacy and safety data will be summarized descriptive for subjects who entered extension and for all subjects who have been treated in the study. No formal statistical inference will be performed.

#### 4.1 Analysis Populations

Extension Safety Population (Safety-EX) and Safety Population are the same defined as in the SAP Part 1.

### 4.2 Handling Dropouts and Missing Data

Missing values in the efficacy and safety parameters will <u>not</u> be imputed. All efficacy and safety will be summarized based on available observed data. Imputation will only be performed on missing or incomplete AE onset date or CM start/stop date. The same imputation algorithm described in SAP Part 1 will be used.

#### 4.3 Definition of Baseline

For subjects who were randomized to FG-3019 arm, the original baseline defined in the Randomized Treatment Period as described in SAP Part 1 will be used. This definition will enable evaluation of long term treatment effect in safety and efficacy parameters.

For subjects who were randomized to placebo arm, baseline in Extension Period will be redefined as last assessment prior to first dose in Extension on Day 1-EX. This will separate the effect of FG-3019 from placebo.

## 4.4 Efficacy Analysis Visit Window

The assessment intervals for the efficacy parameters (PFT, HRCT, and PRO) are the same in the Randomized Treatament Period and Extened Treatment Period, the same windowing rules described in SAP Part 1 will be used.

#### 4.5 General Layout

For subjects who have been treated in extension, all safety and efficacy data, including both the Randomized Treatment Period and Extended Treatment Period, will be summarized descriptively by scheduled visit. All data will be presented in data listings.

#### 5 STATISTICAL ANALYSES

#### 5.1 Subject Disposition

The number of subjects in each study population will be summarized. The number of subjects who completed or discontinued the study as well as the reasons for early discontinuation will be summarized for subjects entered extension.

Subject who discontinued the study prematurely and the reasons will be listed.

#### **5.2** Protocol Deviations

Protocol deviations occurred in the extension period will be summarized and presented in data listing for subjects treated in extension.

## 5.3 Demographic and Baseline Characteristics

Demographics and baseline characteristics will be summarized and presented in data listing as described in Section 4.5.

## 5.4 Summary of Prior and Concomitant Medications

Concomitant medications and non-drug therapies administered during the study will be summarized by study period.

All medications and non-drug therapies will be presented in data listings for subjects treated in extension.

#### 5.5 Summary of Study Drug Exposure and Treatment Compliance

Duration in days from first dose to last dose, number of doses, and dose amount in mg will be summarized and presented in data listing as described in Section 4.5.

### 5.6 Summary of the Efficacy Data in the Extension Period

Efficacy parameters, including change from baseline in FVCpp, FVC (L), HRCT fibrosis score, and SGRQ total and domain scores, are summarized descriptively at each scheduled visit for subjects who have been treated in extension.

#### 5.7 Summary of Safety Data in the Extension Period and Overall Study

#### 5.7.1 Summary of Treatment Emergent Adverse Events and Mortality

TEAE and mortality will be summarized for subjects who entered extension.

#### 5.7.2 Summary of Other Safety Data

Other safety data including central laboratory data, vital signs, ECG, and physical examination will be summarized descriptively by visit for subjects who have received extended treatment.

## 6 CHANGES FROM THE PROTOCOL

• As documented in Note-To-File dated 05DEC2017 biomarker samples collected at Week 24 (pre-dose) and Week 48 at each extension year, are used to evaluate trough level of FG-3019 concentraction.

## APPENDIX. GENERAL SPECIFICATIONS FOR SUBMISSION DATA

## 1. Study Data Tabulation Model (SDTM)

A new set of SDTM datasets, containing the entire study data, will be created. The set of SDTM datasets created for the Randomized Treatment Period is a subset of this set for the entire study.

 Table A.
 Study Data Tabulation Model Datasets (SDTM)

| SDTM<br>Domain | SDTM Domain<br>Description | SDTM Domain<br>Structure | General<br>Observation<br>Class | Source<br>Data Used | Key Variables |
|---|---|---|---|---|---|
| AE | Adverse Events | One record per<br>adverse event per<br>subject | Events | AE | STUDYID,<br>USUBJID,<br>AESTDTC,<br>AEDECOD,<br>AESPID |
| СМ | Concomitant<br>Medications | One record per recorded medication occurrence per subject | Interventions | CM, CMIPF | STUDYID,<br>USUBJID,<br>CMCAT,<br>CMSPID,<br>CMTRT,<br>CMSTDTC |
| DD | Death Details | One record per subject | Findings | DTH | STUDYID,<br>USUBJID,<br>DDTESTCD |
| DM | Demographics | One record per subject | Special<br>Purpose<br>Domains | DM, EX,<br>ICF, DTH,<br>SITE_INV | STUDYID,<br>USUBJID |
| DS | Disposition | one record per disposition status or protocol milestone per subject | | DS, ICF,<br>DTH, EX | STUDYID,<br>USUBJID,<br>DSSTDTC,<br>DSDECOD,<br>DSSPID,<br>EPOCH |
| DV | Protocol<br>Deviations | One record per protocol deviations per subject | Events | DV | STUDYID,<br>USUBJID,<br>DVTERM |
| EC | Exposure as<br>Collected | One record per<br>protocol-specified<br>study treatment per<br>collected-dosing<br>interval per subject | Interventions | EX | STUDYID,<br>USUBJID,<br>ECTRT,<br>ECSTDTC,<br>ECGRPID |
| EG | ECG Test Results | One record per ECG | Findings | EG | STUDYID, |

| | | observation per visit<br>per subject | | | USUBJID,<br>EGTESTCD,<br>VISITNUM |
|---|---|---|---|---|---|
| EX | Exposure | One record per<br>constant dosing<br>interval per subject | Interventions | EX | STUDYID,<br>USUBJID,<br>EXTRT,<br>EXSTDTC |
| IE | Inclusion/Exclusi<br>on Criteria Not<br>Met | One record per inclusion/exclusion criterion not met per subject | Findings | IE | STUDYID,<br>USUBJID,<br>IETESTCD |
| LB | Laboratory Test<br>Results | One record per lab<br>test per specimen<br>per method per<br>LOINC code per<br>reason not done per<br>visit per subject | Findings | eDT LB,<br>RAND,<br>LBC,<br>LBPREG | STUDYID,<br>USUBJID,<br>LBCAT,<br>LBTESTCD,<br>VISITNUM,<br>LBMETHOD,<br>LBREASND,<br>LBLOINC |
| мн | Medical History | One record per<br>medical history<br>event per time<br>interval per subject | Events | МН | STUDYID,<br>USUBJID,<br>MHSPID,<br>MHDECOD,<br>MHSTDTC,<br>MHENDTC |
| PC | Pharmacokinetic<br>Concentrations | One record per time-<br>point concentration<br>or sample<br>characteristic per<br>analyte per subject | Findings | Source documents, PKC | STUDYID,<br>USUBJID,<br>PCTESTCD,<br>VISITNUM,<br>PCTPTNUM |
| PE | Physical<br>Examination | One record per body<br>system or<br>abnormality per visit<br>per subject | Findings | PE | STUDYID,<br>USUBJID,<br>PETESTCD,<br>VISITNUM |
| PP | Pharmacokinetic<br>Parameters | One record per PK parameter per time-concentration profile per modeling method per subject | Findings | Source documents | STUDYID,<br>USUBJID,<br>PPTESTCD,<br>PPCAT,<br>VISITNUM,<br>PPTPTREF |
| PR | Procedures | One record per<br>recorded procedure<br>per occurrence per<br>subject | Interventions | NDT, OU | STUDYID,<br>USUBJID,<br>PRCAT,<br>PRTRT,<br>PRSPID |

| QS | Questionnaires | Questionnaires One record per question per questionnaire per visit per subject | | SGRQ,<br>UCSD | STUDYID,<br>USUBJID,<br>QSTESTCD,<br>VISITNUM |
|---|---|---|---|---|---|
| SC | Subject<br>Characteristics | One record per<br>characteristic per<br>subject | Findings | DM | STUDYID,<br>USUBJID,<br>SCTESTCD |
| SE | Subject Elements | One record per<br>actual Element per<br>subject | Special<br>Purpose<br>Domains | SDTM.DM,<br>SDTM.EX,<br>SDTM.DS,<br>SDTM.SV | STUDYID,<br>USUBJID,<br>TAETORD,<br>SESTDTC |
| SU | Substance Use | One record per<br>substance type per<br>subject | Intervention | SUTOB | STUDYID,<br>USUBJID,<br>SUTRT |
| sv | Subject Visits | One record per<br>actual visit per<br>subject | Special<br>Purpose<br>Domains | All datasets including visits | STUDYID,<br>USUBJID,<br>VISITNUM |
| ТА | Trial Arms | One record per<br>planned Element per<br>Arm | Trial Design | N/A | STUDYID,<br>ARMCD,<br>TAETORD |
| TE | Trial Elements | One record per planned Element | Trial Design | N/A | STUDYID,<br>ETCD |
| TI | Trial<br>Inclusion/Exclusi<br>on Criteria | One record per I/E<br>criterion per<br>protocol criteria<br>version | Trial Design | N/A | STUDYID,<br>TIVERS,<br>IETESTCD |
| TS | Trial Summary | One record per Trial<br>Summary parameter<br>per occurrence | Trial Design | N/A | STUDYID,<br>TSPARMCD,<br>TSSEQ |
| TV | Trial Visits | One record per<br>planned Visit per<br>Arm | Trial Design | N/A | STUDYID,<br>VISITNUM,<br>ARMCD |
| VS | Vital Signs | One record per vital<br>sign measurement<br>per time point per<br>visit per subject | Findings | VS, SC | STUDYID,<br>USUBJID,<br>VSTESTCD,<br>VISITNUM,<br>VSDTC |
| ZH | High Resolution<br>Computed<br>Tomography | One record per<br>examination per<br>location per time<br>point per visit per<br>subject | Findings | HRCT,<br>TEXTCAD,<br>TEXTVIS,<br>IMQUAL | STUDYID,<br>USUBJID,<br>ZHCAT,<br>ZHTESTCD,<br>VISITNUM,<br>ZHDTC, |

| | | | | | ZHLOC,<br>ZHEVAL |
|---|---|---|---|---|---|
| ZI | IPF Confirmation | One record per IPF<br>Confirmation per<br>test per subject | Findings | IPFD | STUDYID,<br>USUBJID,<br>ZITESTCD |
| ZP | Pulmonary<br>Function Tests | One record per test<br>per time point per<br>visit per result per<br>subject | Findings | eDT PFT,<br>RAND, ZP,<br>MHPFT | STUDYID,<br>USUBJID,<br>ZPCAT,<br>ZPTESTCD,<br>VISITNUM,<br>ZPDTC,<br>ZPORRES |

# 2 Analysis Data Model (ADaM)

A new set of ADaM datasets will be created to fit the required analyses for SAP Part 2.

Table B. Analysis Data Model (ADaM)

| Dataset | Description | Structure | Keys |
|---|---|---|---|
| ADSL | Subject-Level<br>Analysis Dataset | One record per subject | STUDYID, SUBJID |
| ADAE | Analysis Dataset<br>Adverse Events | One record per subject per adverse event | STUDYID, SUBJID,<br>AESTDTC,<br>AEDECOD, AESPID |
| ADCM | Analysis Dataset<br>Concomitant<br>Medications | One record per subject per recorded medication occurrence | STUDYID, SUBJID,<br>CMCAT, CMSPID,<br>CMTRT, CMSTDTC |
| ADDD | Analysis Dataset<br>Death | One record per subject per paramter | STUDYID SUBJID<br>PARAMCD |
| ADEG | Analysis Dataset for ECG Test Results | One record per subject per visit | STUDYID, SUBJID,<br>PARAMCD,<br>AVISITN, ADT |
| ADEX | Analysis Dataset<br>Exposure | One record per subject per parameter per visit | STUDYID, SUBJID,<br>PARAMCD, AVISITN |
| ADHRCT | Analysis Dataset<br>HRCT | One record per subject<br>per measurement method<br>per Lung Lobe per<br>parameter per visit | STUDYID, SUBJID,<br>PARAMCD,<br>AVISITN,<br>DTYPE ALOC |
| ADLB | Analysis Dataset<br>Laboratory Test | One record per subject per category per | STUDYID, SUBJID,<br>PARCAT1, |

| | Results | parameter per visit per<br>normal range per result | PARCAT2,<br>PARAMCD,<br>AVISITN, ANRHI,<br>AVAL |
|---|---|---|---|
| ADMH | Analysis Dataset<br>Medical History | One record per subject<br>per medical history per<br>time interval of medical<br>history | STUDYID, SUBJID,<br>MHSPID,<br>MHDECOD,<br>MHSTDTC,<br>MHENDTC |
| ADPC | Analysis Dataset<br>PK Concentrations | One record per subject per visit per time point per parameter | STUDYID, SUBJID,<br>AVISITN, ATPTN,<br>PARAMCD |
| ADPE | Analysis Dataset<br>Physical<br>Examination | One record per subject per parameter per visit | STUDYID, SUBJID,<br>AVISITN, PARAMCD |
| ADPF | Analysis Dataset<br>Pulmonary Function<br>Tests | One record per subject per parameter per time point per visit | USUBJID, SUBJID,<br>PARAMCD,<br>AVISITN, DTYPE,<br>ADT, ATM |
| ADPP | Analysis Dataset<br>Pharmacokinetic<br>Parameters | One record per subject per parameter per visit | STUDYID, SUBJID,<br>AVISITN,<br>PARAMCD |
| ADPR | Analysis Dataset<br>Procedures | One record per recorded procedure per occurrence per subject | STUDYID, SUBJID,<br>PRTRT, PRSPID |
| ADQS | Analysis Dataset for<br>Questionnaire | One record per subject per category per parameter per visit | STUDYID, SUBJID,<br>PARCAT1,<br>PARAMCD,<br>AVISITN, VISITNUM |
| ADTTE | Analysis Dataset<br>Time-to-Event | One record per subject per parameter | STUDYID, SUBJID,<br>PARAMCD |
| ADVS | Analysis Dataset<br>Vital Signs | One record per subject<br>per parameter per time<br>point per visit | STUDYID, SUBJID,<br>PARAMCD,<br>AVISITN, DTYPE,<br>ADT, ATM, ATPTN |